CLINICAL TRIAL: NCT00939770
Title: A Phase 1/2 Study of Crizotinib, an Oral Small Molecule Inhibitor of Anaplastic Lymphoma Kinase (ALK) and C-Met, in Children With Relapsed/Refractory Solid Tumors and Anaplastic Large Cell Lymphoma
Brief Title: Crizotinib in Treating Younger Patients With Relapsed or Refractory Solid Tumors or Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0912; NCI-2011-01937 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P10666; COG-ADVL0912; CDR0000647587; ADVL0912 (Other: Pediatric Early Phase Clinical Trial Network); ADVL0912 (Other: CTEP); UM1CA097452 (NIH); NCT01182896 (obsolete NCT alias)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Neuroblastoma; Refractory Anaplastic Large Cell Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Neuroblastoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Neuroblastoma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (crizotinib) (Experimental): Patients receive crizotinib PO BID on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Crizotinib — Given PO
  Other Names: MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066; PF-2341066; Xalkori
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase 1/2 trial the studies side effects and best dose of crizotinib and to see how well it works in treating young patients with solid tumors or anaplastic large cell lymphoma that has returned after a period of improvement or does not respond to treatment. Crizotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. (Phase 1 completed 2/15/13)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and recommend a Phase 2 dose of Crizotinib administered orally twice daily to children with relapsed/refractory solid tumors and anaplastic large cell lymphoma (ALCL). (completed 2/15/13) II. To define and describe the toxicities of Crizotinib administered on this schedule.

III. To characterize the pharmacokinetics of Crizotinib in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the anti-tumor activity of Crizotinib within the confines of a Phase 1 study. (completed 2/15/13) II. To obtain initial Phase 2 data on the anti-tumor activity of Crizotinib in children with relapsed/refractory neuroblastoma and ALCL.

III. To preliminarily examine the relationship between anaplastic lymphoma kinase (ALK) status (e.g, the presence of a mutation, duplication, amplification, and/or translocation) in patients with neuroblastoma (NB) or ALCL and response to Crizotinib.

IV. To preliminarily examine the relationship between minimal residual disease (MRD) status and clinical response to Crizotinib in patients with ALCL.

V. To use a questionnaire to gather preliminary information on the palatability of the oral solution formulation of Crizotinib.

VI. To evaluate for potential alterations in bone growth in pediatric patients.

OUTLINE: This is a phase 1 dose-escalation study (completed 2/15/13) followed by a phase 2 study.

Patients receive crizotinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving the formulated capsules must have a body surface area (BSA) >= 0.63 m^2 at the time of study enrollment
* Patients must have had histologic verification of malignancy at original diagnosis or relapse
* * Phase 1 (Part A1) - COMPLETE: Patients with relapsed or refractory solid tumors or anaplastic large cell lymphoma (excluding patients with primary or metastatic central nervous system [CNS] tumors or patients with primary cutaneous ALCL)
* * Phase 1 (Part A2) - COMPLETE: Patients with confirmed ALK fusion proteins, ALK mutations, ALK amplification (defined as greater than 4-fold increase in the ALK signal number as compared to reference signal number on chromosome 2q arm) or MET proto-oncogene, receptor tyrosine kinase (MET) mutation or amplification; testing to confirm the presence of ALK fusion proteins, ALK mutations, ALK amplification or evidence of MET mutation or amplification for eligibility purposes must be performed as a Clinical Laboratory Improvement Act (CLIA)-certified assay; ALK immunohistochemistry can be used as a surrogate for fluorescent in situ hybridization (FISH) for patients with inflammatory myofibroblastic tumors (IMT) or ALCL
* ** Note: Evidence for MET mutation or amplification is defined as:

  * Positive for c-Met amplification by FISH; or
  * Positive for known c-Met kinase domain activating mutations including V1110L, H1112L, H1112Y, H1124D, M1149T, T1191I, V1206L, L1213V, V1238I, M1268T, P1009S, T1010I, R988C, V941L, but excluding Y1248C, Y1248H, Y1248D, and Y1253D; or
  * Chromosomal translocations that lead to altered transcriptional regulation of c-Met and/or hepatocyte growth factor (HGF) including metastatic alveolar soft part sarcoma, clear cell sarcoma, rhabdomyosarcoma, or translocation associated renal cell carcinoma)
* * Phase 1 (Part A3) - COMPLETE: Patients with relapsed or refractory neuroblastoma, with or without bone marrow involvement, who are not eligible for Part A1 or A2 or cannot enroll on Part A1 because of stratum suspension or lack of available slots (these patients will be enrolled at one dose level below the dose level at which patients on Part A1 are actively enrolling)
* * Phase 2 (Part B): Patients with ALK+ relapsed or refractory neuroblastoma
* * Phase 2 (Part C): Patients with ALK+ relapsed or refractory ALCL (excluding patients with primary cutaneous ALCL)
* * Phase 2 (Part A2): Patients with diagnoses other than neuroblastoma or ALCL with confirmed ALK fusion proteins, ALK mutations, ALK amplification (defined as greater than 4-fold increase in the ALK signal number as compared to reference signal number on chromosome 2q arm) or MET mutation or amplification; testing to confirm the presence of ALK fusion proteins, ALK mutations, ALK amplification or evidence of MET mutation or amplification for eligibility purposes must be performed as a CLIA-certified assay; ALK immunohistochemistry can be used as a surrogate for FISH for patients with IMT
* Disease status:

  * Phase 1 (Part A): Patients must have either measurable and/or evaluable disease
  * Phase 2 (Part B): Patients with neuroblastoma must have proven ALK+ disease with either measurable and/or evaluable disease as indicated below:

    * Measurable tumor on magnetic resonance imaging (MRI), computed tomography (CT) scan or X-ray obtained within 2 weeks prior to study enrollment
    * Evaluable tumor by meta-iodobenzyl guanidine I 123 (MIBG) scan and/or bone marrow involvement with tumor cells seen on routine morphology
  * Phase 2 (Part C): Patients must have proven ALK+ disease with either measurable or evaluable disease
* Performance level: Karnofsky >= 50 for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age); Note: patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy:

  * Myelosuppressive chemotherapy:

    * Solid tumors: Patients with solid tumors must not have received chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
    * Lymphoma: Patients with lymphoma who relapse during standard maintenance therapy are eligible at time of relapse; for patients with ALCL who relapse while they are receiving cytotoxic therapy, at least 14 days must have elapsed since the completion of cytotoxic therapy; Note: cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of Crizotinib
* At least 7 days since the completion of therapy with a growth factor
* At least 7 days since the completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 7 days or 3 half-lives, whichever is longer, must have elapsed since prior treatment with a monoclonal antibody
* >= 2 weeks (wks) for local palliative radiation therapy (XRT) (small port); >= 6 weeks must have elapsed since treatment with therapeutic doses of MIBG; >= 6 months must have elapsed if prior total body irradiation (TBI), craniospinal XRT or >= 50% radiation of pelvis; >= 6 wks must have elapsed if other substantial bone marrow (BM) radiation
* Bone marrow/stem cell transplant or infusion without TBI:

  * Part A1 or Part C: No evidence of active graft vs host disease and >= 3 months must have elapsed since stem cell transplant or infusion
  * Part A2, Part A3, or Part B: No evidence of active graft vs host disease and >= 6 weeks must have elapsed since stem cell transplant or infusion
* At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
* Patients must not have received prior therapy with Crizotinib
* Patients on Part A1 or Part C of the study:

  * For patients with solid tumors or ALCL without bone marrow involvement:

    * Peripheral absolute neutrophil count (ANC) >= 1,000/mm^3
    * Platelet count >= 75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
    * Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
  * Patients with known bone marrow metastatic disease:

    * Peripheral absolute neutrophil count (ANC) >= 750/mm^3
    * Platelet count >= 25,000/mm^3 (may receive platelet transfusions)
    * Hemoglobin >= 8.0 g/dL (may receive RBC transfusions)
    * Not known to be refractory to RBC or platelet transfusions Transfusions are permitted to meet both the platelet and hemoglobin criteria; Note: patients with known bone marrow metastatic disease are not evaluable for hematological toxicity for the purposes of dose escalation
* Patients eligible for Part A2, Part A3, or Part B of the study must meet the hematologic criteria below for enrollment:

  * Peripheral absolute neutrophil count (ANC) >= 750/mm^3
  * Platelet count >= 25,000/mm^3 (may receive platelet transfusions)
  * Hemoglobin >= 8.0 g/dL (may receive RBC transfusions)
  * Not known to be refractory to red cell or platelet transfusions Transfusions are permitted to meet both the platelet and hemoglobin criteria
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male), 1.4 mg/dL (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Corrected QT interval (QTc) =< 480 msec
* All patients and/or their parents or legal guardians must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Patients taking the capsule formulation must be able to swallow capsules; feeding tube administration is allowed for patients receiving the oral solution (OS)

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the prior 7 days are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents, with the exception of hydroxyurea for patients with ALCL, are not eligible
* As Crizotinib is an inhibitor of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), patients chronically receiving medications known to be metabolized by CYP3A4 and with narrow therapeutic indices including pimozide, aripiprazole, triazolam, ergotamine and halofantrine are not eligible; the topical use of these medications (if applicable) is allowed
* Patients chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment, including but not limited to, ketoconazole, itraconazole, miconazole, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, amprenavir, delavirdine, nefazodone, diltiazem, verapamil, and grapefruit juice are not eligible; the topical use of these medications (if applicable), e.g. 2% ketoconazole cream, is allowed
* Patients chronically receiving drugs that are known potent CYP3A4 inducers within 12 days prior to study enrollment, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, tipranavir, ritonavir, and St. John's wort are not eligible; the topical use of these medications (if applicable) is allowed
* Patients with known interstitial fibrosis or interstitial lung disease are not eligible
* Patients with a known history of myocardial infarction or cerebrovascular accident are not eligible
* Patients with central nervous system (CNS) tumors or known CNS metastases are not eligible; patients with a history of CNS metastases that have been surgically resected are eligible only if the baseline evaluation shows no evidence of current CNS metastases; patients with any evidence of CNS metastases on baseline evaluation are not eligible, regardless of whether the lesions have been previously treated and/or appear stable
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael P Mosse, Principal Investigator — COG Phase I Consortium
Locations (28):
- United States (27):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Foster JH, Voss SD, Hall DC, Minard CG, Balis FM, Wilner K, Berg SL, Fox E, Adamson PC, Blaney SM, Weigel BJ, Mosse YP. Activity of Crizotinib in Patients with ALK-Aberrant Relapsed/Refractory Neuroblastoma: A Children's Oncology Group Study (ADVL0912). Clin Cancer Res. 2021 Jul 1;27(13):3543-3548. doi: 10.1158/1078-0432.CCR-20-4224. Epub 2021 Feb 10. PMID 33568345
- [Derived] Balis FM, Thompson PA, Mosse YP, Blaney SM, Minard CG, Weigel BJ, Fox E. First-dose and steady-state pharmacokinetics of orally administered crizotinib in children with solid tumors: a report on ADVL0912 from the Children's Oncology Group Phase 1/Pilot Consortium. Cancer Chemother Pharmacol. 2017 Jan;79(1):181-187. doi: 10.1007/s00280-016-3220-6. Epub 2016 Dec 28. PMID 28032129
- [Derived] Mosse YP, Lim MS, Voss SD, Wilner K, Ruffner K, Laliberte J, Rolland D, Balis FM, Maris JM, Weigel BJ, Ingle AM, Ahern C, Adamson PC, Blaney SM. Safety and activity of crizotinib for paediatric patients with refractory solid tumours or anaplastic large-cell lymphoma: a Children's Oncology Group phase 1 consortium study. Lancet Oncol. 2013 May;14(6):472-80. doi: 10.1016/S1470-2045(13)70095-0. Epub 2013 Apr 16. PMID 23598171

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID; Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID: Part A1: Patients with relapsed/refractory solid tumors or anaplastic large cell lymphoma (ALCL) Part A2: Patients with recurrent/refractory malignancies who have confirmed ALK fusion proteins, ALK mutations, ALK amplification or evidence for MET mutation or amplification. Once Parts B and C are open to accrual, patients who are not eligible for either Part should enroll on Part A2, Part A3: Patients with recurrent/refractory neuroblastoma, who are not eligible for Part A1 or A2 or who cannot enroll on Part A1 because of stratum suspension or lack of available slots.
- Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID: Part B: Patients with ALK+ relapsed/refractory neuroblastoma
- Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID: Part C: Patients with ALK+ relapsed/refractory ALCL
Period: Overall Study
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID
Started | 6 | 8 | 23 | 12 | 38 | 11 | 14 | 10
Completed | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Not Completed | 5 | 8 | 20 | 11 | 37 | 11 | 14 | 10
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 6 | 2 | 1 | 1
Not completed — Lack of Efficacy | 4 | 6 | 13 | 9 | 16 | 8 | 11 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 7 | 1 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 5 | 2 | 6 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase 1:Part A: PF-02341066 130 mg/m²/Dose BID; Phase 1:Part A: PF-02341066 165 mg/m²/Dose BID; Phase 1:Part A: PF-02341066 215 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 280 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 365 mg/m²/Dose BID: Part A1: Patients with relapsed/refractory solid tumors or anaplastic large cell lymphoma (ALCL) Part A2: Patients with recurrent/refractory malignancies who have confirmed ALK fusion proteins, ALK mutations, ALK amplification or evidence for MET mutation or amplification. Once Parts B and C are open to accrual, patients who are not eligible for either Part should enroll on Part A2, Part A3: Patients with recurrent/refractory neuroblastoma, who are not eligible for Part A1 or A2 or who cannot enroll on Part A1 because of stratum suspension or lack of available slots.
- Phase 2: Part B: PF-02341066 280 mg/m²/Dose BID: Part B: Patients with ALK+ relapsed/refractory neuroblastoma
- Phase 2: Part C: PF-02341066 280 mg/m²/Dose BID: Part C: Patients with ALK+ relapsed/refractory ALCL
- Total: Total of all reporting groups
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1:Part A: PF-02341066 130 mg/m²/Dose BID | Phase 1:Part A: PF-02341066 165 mg/m²/Dose BID | Phase 1:Part A: PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 280 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m²/Dose BID | Phase 2: Part B: PF-02341066 280 mg/m²/Dose BID | Phase 2: Part C: PF-02341066 280 mg/m²/Dose BID | Total
Number analyzed (Participants) | 6 | 8 | 23 | 12 | 38 | 11 | 14 | 10 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 21 | 11 | 34 | 10 | 14 | 10 | 113
  Between 18 and 65 years | 0 | 1 | 2 | 1 | 4 | 1 | 0 | 0 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8.5 [5 to 12] | 12 [6 to 20] | 8 [1 to 21] | 11.5 [3 to 20] | 9 [1 to 21] | 10 [2 to 20] | 5.5 [3 to 14] | 9.5 [6 to 15] | 9 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 9 | 6 | 25 | 5 | 8 | 2 | 60
  Male | 4 | 5 | 14 | 6 | 13 | 6 | 6 | 8 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 6 | 2 | 1 | 1 | 13
  Not Hispanic or Latino | 5 | 8 | 21 | 7 | 28 | 8 | 13 | 8 | 98
  Unknown or Not Reported | 1 | 0 | 1 | 3 | 4 | 1 | 0 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 5 | 1 | 1 | 3 | 11
  White | 5 | 6 | 19 | 8 | 25 | 8 | 12 | 4 | 87
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 4 | 7 | 1 | 0 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose and Recommended Phase 2 Dose of Crizotinib
Description: The descriptions and grading scales found in the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for adverse event (AE) reporting. The MTD/RP2D is defined as the maximum dose at which fewer than one-third of patients experience dose limiting toxicity.
Time Frame: 28 days
Population: Phase 1 patients
Measure: Number; unit: mg/m²/dose BID
Groups:
- Part A: Part A1: Patients with relapsed/refractory solid tumors or anaplastic large cell lymphoma (ALCL) Part A2: Patients with recurrent/refractory malignancies who have confirmed ALK fusion proteins, ALK mutations, ALK amplification or evidence for MET mutation or amplification. Once Parts B and C are open to accrual, patients who are not eligible for either Part should enroll on Part A2, Part A3: Patients with recurrent/refractory neuroblastoma, who are not eligible for Part A1 or A2 or who cannot enroll on Part A1 because of stratum suspension or lack of available slots.
Arm/Group | Part A
Number analyzed (Participants) | 98
mg/m²/dose BID | 280

2. Primary Outcome: Number of Participants With Toxicities of Crizotinib
Description: The descriptions and grading scales found in the revised NCI CTCAE version 4.0 will be utilized for AE reporting.
Time Frame: Up to 30 days post-treatment
Population: All patients included in analysis
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Part A:PF-02341066 130 mg/m²/Dose BID; Phase 1: Part A:PF-02341066 165 mg/m²/Dose BID; Phase 1: Part A:PF-02341066 215 mg/m²/Dose BID; Phase 1: Part A:PF-02341066 280 mg/m²/Dose BID; Phase 1: Part A: PF-02341066 365 mg/m²/Dose BID: Part A1: Patients with relapsed/refractory solid tumors or anaplastic large cell lymphoma (ALCL) Part A2: Patients with recurrent/refractory malignancies who have confirmed ALK fusion proteins, ALK mutations, ALK amplification or evidence for MET mutation or amplification. Once Parts B and C are open to accrual, patients who are not eligible for either Part should enroll on Part A2, Part A3: Patients with recurrent/refractory neuroblastoma, who are not eligible for Part A1 or A2 or who cannot enroll on Part A1 because of stratum suspension or lack of available slots.
- Phase 2:Part C: PF-02341066 280 mg/m2/Dose BID: Part C: Patients with ALK+ relapsed/refractory ALCL
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1: Part A:PF-02341066 130 mg/m²/Dose BID | Phase 1: Part A:PF-02341066 165 mg/m²/Dose BID | Phase 1: Part A:PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A:PF-02341066 280 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m²/Dose BID | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID | Phase 2:Part C: PF-02341066 280 mg/m2/Dose BID
Number analyzed (Participants) | 6 | 8 | 23 | 12 | 38 | 11 | 14 | 10
Participants | 6 | 7 | 23 | 11 | 38 | 11 | 14 | 10

3. Primary Outcome: Steady State C Max of Crizotinib
Description: Mean with standard deviation of peak of serum concentration curve at steady state by dose level.
Time Frame: Cycle 1 (day 15- 28) pre-dose, 1, 2,4, 6-8 hours post dose
Population: Steady state PK sampling was not performed during enrollment on dose level 1 or 2. In Phase 2, PK was optional and for those who consented data is included with dose level 5. Steady state PK samples were obtained on a day between day 15 and 28 of cycle 1, pre-dose, 1, 2, 4, 6-8 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Level 3: PF-02341066 165 mg/m²/dose BID
- Dose Level 4: PF-02341066 215 mg/m²/dose BID
- Dose Level 5: PF-02341066 280 mg/m²/dose BID
- Dose Level 6: PF-02341066 365 mg/m²/dose BID
Arm/Group | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 1 | 5 | 36 | 6
ng/mL | 294 (0) | 601 (118) | 717 (201) | 972 (210)

4. Primary Outcome: Steady State C Average of Crizotinib
Description: Mean with standard deviation of average serum concentration curve at steady state by dose level.
Time Frame: Cycle 1 (day 15-28) pre-dose, 1, 2, 4, 6-8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 1 | 5 | 36 | 6
ng/mL | 246 (0) | 469 (114) | 582 (173) | 731 (228)

5. Primary Outcome: Steady State AUC of Crizotinib
Description: Mean with standard deviation of area under the serum concentration curve at steady state by dose level.
Time Frame: Cycle 1 (day 15-28) pre-dose, 1, 2, 4, 6-8 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ng•h/mL
Arm/Group | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 1 | 5 | 36 | 6
ng•h/mL | 2950 (0) | 5630 (1370) | 6990 (2080) | 8770 (2740)

6. Primary Outcome: Steady State Clearance of Crizotinib
Description: Mean with standard deviation of the elimination of crizotinib at steady state by dose level.
Time Frame: Cycle 1 (day 15-28) pre-dose, 1, 2, 4, 6-8 hour post-dose
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mL/min/m2
Arm/Group | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 1 | 5 | 36 | 6
mL/min/m2 | 735 (0) | 652 (159) | 736 (255) | 731 (223)

7. Secondary Outcome: Number of Participants (Relapsed or Refractory Solid Tumors or Anaplastic Large Cell Lymphoma (ALCL))With Response to Crizotinib
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 8 years
Population: Part A Participants with relapsed or refractory solid tumors or anaplastic large cell lymphoma (ALCL)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID
Number analyzed (Participants) | 6 | 8 | 23 | 12 | 38 | 11
Participants | 0 | 0 | 7 | 0 | 19 | 1

8. Secondary Outcome: Number of Participants (Relapsed or Refractory Neuroblastoma or Anaplastic Large Cell Lymphoma (ALCL)) With Response to Crizotinib
Description: as for outcome 7
Time Frame: Up to 8 years
Population: Part B and Part C participants with relapsed or refractory neuroblastoma or anaplastic large cell lymphoma (ALCL)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID
Number analyzed (Participants) | 14 | 10
Participants | 1 | 7

9. Secondary Outcome: Number of Participants With Minimum Residual Disease (MRD)
Description: MRD status will be reported descriptively. The relationship between MRD status and clinical response to treatment will be examined in children with ALCL.
Time Frame: Up to 8 years
Population: MRD Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID
Number analyzed (Participants) | 6 | 8 | 23 | 12 | 38 | 11 | 14 | 10
Participants | 0 | 0 | 5 | 0 | 9 | 0 | 0 | 10

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 3/23 | 2/12 | 2/38 | 1/11 | 1/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/8 | 18/23 | 10/12 | 33/38 | 11/11 | 13/14 | 10/10
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 23/23 | 12/12 | 38/38 | 11/11 | 14/14 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID (N=6) | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID (N=8) | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID (N=23) | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID (N=12) | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID (N=38) | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID (N=11) | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID (N=14) | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abducens nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 1 | 5 | 0 | 4 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0 | 1 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aortic injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 1
Fever (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 3 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 2 | 0 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 5 | 1 | 2 | 0 | 1 | 1
Infective myositis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
IVth nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 3 | 7 | 2 | 9 | 1 | 6 | 5
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 3 | 10 | 6 | 18 | 7 | 10 | 10
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 4 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 2 | 3 | 1 | 7 | 0 | 4 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 2 | 3 | 3 | 9 | 1 | 4 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Part A: PF-02341066 100 mg/m²/Dose BID (N=6) | Phase 1: Part A: PF-02341066 130 mg/m²/Dose BID (N=8) | Phase 1: Part A: PF-02341066 165 mg/m²/Dose BID (N=23) | Phase 1: Part A: PF-02341066 215 mg/m²/Dose BID (N=12) | Phase 1: Part A: PF-02341066 280 mg/m2/Dose BID (N=38) | Phase 1: Part A: PF-02341066 365 mg/m2/Dose BID (N=11) | Phase 2: Part B: PF-02341066 280 mg/m2/Dose BID (N=14) | Phase 2: Part C: PF-02341066 280 mg/m2/Dose BID (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 5 | 1 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 13 | 2 | 18 | 3 | 7 | 2
Abducens nerve disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Accessory nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 3 | 0 | 2 | 2 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 8 | 0 | 4 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 3 | 20 | 11 | 33 | 8 | 12 | 9
Alkaline phosphatase increased (Investigations) | 0 | 2 | 9 | 5 | 12 | 2 | 2 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 8 | 1 | 10 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 6 | 1 | 5 | 4 | 8 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 6 | 20 | 8 | 33 | 11 | 13 | 7
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 11 | 6 | 19 | 7 | 8 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 4 | 3 | 4 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 7 | 2 | 1 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 21 | 11 | 33 | 11 | 14 | 8
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3 | 5 | 4 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1
Blood antidiuretic hormone abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 2 | 6 | 3 | 15 | 2 | 1 | 3
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1 | 3 | 2 | 2 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 6 | 1 | 2 | 0 | 1 | 1
Cholesterol high (Investigations) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 9 | 6 | 14 | 3 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 16 | 5 | 24 | 3 | 7 | 4
CPK increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 5 | 2 | 15 | 5 | 16 | 6 | 9 | 3
Cushingoid (Endocrine disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3 | 1 | 2 | 2 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 3 | 2 | 1 | 2 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 15 | 6 | 25 | 9 | 11 | 10
Dizziness (Nervous system disorders) | 0 | 0 | 7 | 2 | 7 | 2 | 2 | 2
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 1 | 4 | 2 | 2 | 2
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 2 | 5 | 2 | 1 | 4
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 2 | 4 | 1 | 2 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1
Edema face (General disorders) | 0 | 0 | 2 | 1 | 3 | 1 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 4 | 2 | 8 | 0 | 0 | 1
Edema trunk (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1 | 1 | 4 | 1 | 1 | 2
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Esophageal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Euphoria (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 2 | 1 | 7 | 2 | 10 | 3 | 4 | 7
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 2
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 17 | 9 | 24 | 8 | 9 | 6
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 13 | 4 | 19 | 2 | 9 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 3 | 0 | 1 | 1
Floaters (Eye disorders) | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 2
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 4 | 0 | 2 | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 0
Gait disturbance (General disorders) | 2 | 1 | 2 | 1 | 4 | 1 | 4 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 3
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 1 | 2 | 6 | 1 | 9 | 4 | 4 | 2
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Gum infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 14 | 7 | 12 | 3 | 4 | 6
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 5 | 1 | 4 | 0 | 4 | 1
Hemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hemoglobinuria (Renal and urinary disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2 | 16 | 6 | 23 | 5 | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 8 | 3 | 10 | 0 | 5 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 5 | 4 | 13 | 3 | 2 | 5
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 5 | 1 | 3 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 9 | 0 | 10 | 0 | 3 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 4 | 18 | 5 | 30 | 5 | 11 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4 | 18 | 8 | 21 | 5 | 6 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1 | 14 | 4 | 3 | 4
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4 | 10 | 5 | 12 | 4 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 9 | 0 | 5 | 2 | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | 11 | 0 | 13 | 3 | 5 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0 | 8 | 6 | 10 | 5 | 6 | 2
Hypotension (Vascular disorders) | 2 | 2 | 7 | 2 | 4 | 2 | 3 | 3
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 6 | 1 | 9 | 1 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 3 | 1 | 6 | 0 | 1 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0
IVth nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Lymphedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 6 | 15 | 8 | 22 | 8 | 10 | 3
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 5 | 0 | 1 | 1
Movements involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 1 | 0 | 2 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 4 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1 | 5 | 0 | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 6 | 21 | 9 | 31 | 9 | 10 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 18 | 5 | 25 | 6 | 11 | 5
Non-cardiac chest pain (General disorders) | 0 | 1 | 8 | 3 | 5 | 2 | 0 | 2
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 0
Pain (General disorders) | 2 | 1 | 8 | 2 | 11 | 1 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 8 | 4 | 20 | 4 | 5 | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Papilledema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 3 | 0 | 5 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 3 | 1 | 4 | 2 | 1 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 4 | 0 | 1 | 1 | 2 | 1
Platelet count decreased (Investigations) | 3 | 3 | 12 | 3 | 8 | 1 | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 2 | 1 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4 | 7 | 2 | 6 | 3 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 1 | 7 | 1 | 2 | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 13 | 2 | 8 | 2 | 0 | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 1 | 8 | 0 | 2 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 5 | 1 | 4 | 1 | 2 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 10 | 0 | 4 | 2 | 7 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 9 | 1 | 9 | 1 | 3 | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 4 | 0 | 3 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 2 | 10 | 1 | 3 | 2
Stomach pain (Gastrointestinal disorders) | 2 | 0 | 4 | 0 | 4 | 3 | 0 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 8 | 1 | 7 | 1 | 3 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vagus nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 20 | 9 | 29 | 11 | 13 | 10
Watering eyes (Eye disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 0 | 5 | 0 | 6 | 0 | 3 | 1
Weight loss (Investigations) | 1 | 0 | 5 | 3 | 5 | 1 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 4 | 3 | 20 | 7 | 31 | 10 | 12 | 8
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT00939770/Prot_SAP_ICF_001.pdf